CLINICAL TRIAL: NCT03577041
Title: Medico-economic Evaluation of Anti-VEGF Treatments in the Treatment of naïve Age-related Macular Degeneration (AMD): a Model Adapted to the French Context
Acronym: MEDIAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0009
Record Dates: First submitted 2018-06-04; First posted 2018-07-05 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-02

CONDITIONS: Age-related Macular Degeneration (AMD)
Keywords: Neovascular Age-Related Macular Degeneration; Bevacizumab; Cost-Effective; Quality of life
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Age-related macular degeneration (AMD) is the leading cause of blindness after 50 years in industrialized countries, compromising daily activities and reducing quality of life. And whose treatment is one of the first health expenditures. Since September 2015, Bevacizumab, which does not have marketing authorization in AMD, has been given a temporary recommendation for use. Studies in other countries have shown that bevacizumab is cost-effective in the treatment of AMD compared to other anti-VEGF therapies used.

DETAILED DESCRIPTION:
Numerous clinical trials have shown the effectiveness of Bevacizumab in the treatment of neovascular AMD as well that non-inferiority compared to Ranibizumab in terms of clinical efficacy at 1 year on visual acuity measured by the ETDRS scale of patients with neovascular AMD.

Regarding general tolerance, a recent meta-analysis including a large number of patients did not find any difference in systemic serious adverse reactions, neither any new special signal of tolerance with Bevacizumab. Concerning eye tolerance, there is no evidence of difference significant. Medico-economic analyzes carried out in other countries, as the United States or Brazil, have shown that Bevacizumab is cost-effective compared to Ranibizumab in AMD Neovascular.

The cost-utility analysis of the different methods of care patients with AMD will rely on the construction of a self-centered model built from: data available in natural history literature AMD in the absence of treatment; results of the network meta-analysis comparing effectiveness and tolerance of different strategies to assess; available data on adherence and persistence of treatments; pharmacovigilance data on the occurrence of side effects.

This analysis benefits from two related studies:

* Micro-costing, multicenter study of the preparation of intravitreal injections of Bevacizumab hospital pharmacy.
* Multicenter, prospective evaluation, cross-section, quality of life data and patient cost depending on the level of visual acuity.

According to the recommendations, at the beginning of the treatment, after the diagnosis of neovascular naive AMD, the patient will benefit from a fixed regimen of treatment by intravitreous injection of Bevacizumab or Ranibizumab or Aflibercept renewed every month for 3 months. Before each Intra-vitreous injection, the patient will be reviewed in consultation to collect the occurrence of events adverse reactions related to the injection of one of the three products. After 3 months, the monthly intra-vitreous injections will be left to the appreciation of the investigator.

The follow-up of the patients, during a specialized consultation will be spread out over 6 months according to the rhythm of a consultation by months and then 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Naive neovascular AMD form of retro localization foveal, unilateral or bilateral (one eye per patient will be studied),
* Patients to be treated with intravitreous injections of Bevacizumab or Ranibizumab or Aflibercept,
* Patient using effective contraception if he is of childbearing age
* Patient informed and not having made his opposition to the research,
* Patient under social security scheme.

Exclusion Criteria:

* Previous or current treatment of AMD by intravenous injection of anti-VEGF or surgery dating less than 2 months in the studied eye,
* Contraindications to the taking of Bevacizumab or Ranibizumab or Aflibercept,
* Aphakia in the studied eye,
* Fibrosis or retrofoveolar retinal atrophy of the eye studied,
* Tearing of the pigment epithelium reaching my macula of the studied eye,
* Choroidal neovascularization unrelated to AMD,
* Diabetic retinopathy and / or diabetic maculopathy proven,
* Glycated hemoglobin greater than 12%,
* Known hypersensitivity to pharmaceutical agents used,
* Pregnant or lactating women,
* Severe active intraocular inflammation, or history autoimmune or idiopathic uveitis,
* Active or suspected ocular or periocular infection,
* Intraocular pressure> 25mmHg despite two hypotonizing treatments in eye drops,
* Patient under tutorship or curatorship or private public law.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 50 years of age with a naive neovascular AMD form with a retro-fleeal, unilateral or bilateral location, to be treated with intravitreous injections of Bevacizumab or Ranibizumab or Aflibercept according to the practice of each service
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Cost-utility analysis of the modalities of management of neovascular age-related macular degeneration | 12 months
  Using a probabilistic Markov model

SECONDARY OUTCOMES:
Micro-costing type evaluation of packaging of Intravitreal injections of Bevacizumab in pharmacy hospital. | 12 months
  Costs of packaging of Intravitreal injections of Bevacizumab in pharmacy hospital (flasks of Bevacizumab, materials, personal, infrastructure, conservation)
Quality of life coefficient: HUI 3 questionnaire | 12 months
  Quality of life will be estimated using the HUI 3 questionnaire and corresponding value-set

CONTACTS AND LOCATIONS:
Overall Officials: Sophie BRYSELBOUT, Dr, Study Director — CHU Amiens; Marc MURAINE, Pr, Principal Investigator — CHU Rouen; Xavier ZANLONGHI, Dr, Principal Investigator — Nantes University Hospital; Carl ARNDT, Principal Investigator — Carl
Locations (1):
- CHU Amiens, Amiens, France